CLINICAL TRIAL: NCT03235765
Title: Clinical Validity of Oncogenic Driver Genes Detected From Circulating Tumor DNA in Blood of Lung Cancer Patients
Brief Title: Cancer Panel From Blood of Lung Cancer Patients
Acronym: CAPABLE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: MACROGEN (Other)
Responsible Party: Principal Investigator, Jong-Seok Lee, Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-17-01
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Recurrent
Keywords: NSCLC; Cancer panel; NGS; Actionable mutation; Immune checkpoint inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Cancer panel analysis will be done with patients tumro tissue and ctDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Patients who are diagnosed with metastatic/recurrent non-small cell lung cancer and planned to receive first line chemotherapy
  Interventions: Diagnostic Test: MACROGEN Pan Cancer Panel (Tier 2)
- Cohort B: Patients with recurrent/metastatic non-small cell lung cancer who have been receiving molecular targeted therapy, including immune checkpoint inhibitor, and have tumor shrinkage with the agent.
  Interventions: Diagnostic Test: MACROGEN Pan Cancer Panel (Tier 2)

INTERVENTIONS:
Diagnostic Test: MACROGEN Pan Cancer Panel (Tier 2) — This study will utilize a MACROGEN Pan Cancer Panel (Tier 2), which is a hybrid capture-based NGS assay interrogating the coding regions of 170 cancer-related genes.

SUMMARY:
Molecular profiling of lung cancers using circulating tumor DNA (ctDNA) in the blood of patients is rapidly becoming established as a useful source of information to aid clinical decision-making. This study is aimed to to compare concordance rate between tissue based cancer panel analysis and blood based cancer panel analysis in lung cancer patients (both by NGS technique).

DETAILED DESCRIPTION:
This study is comprised of two cohorts as below:

Cohort A: inoperable, untreated, non-small cell lung cancer patients

Cohort B: non-small cell lung cancer patients who are in the treatment with targeted agents including immune checkpoint inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures, sampling, and analyses
* Pathologically confirmed non-small cell lung cancer
* Male or female, aged at least 20 years
* Matches one of two criteria :

  1. Cohort A: Patients who are diagnosed with metastatic/recurrent non-small cell lung cancer and planned to receive first line chemotherapy
  2. Cohort B: Patients with recurrent/metastatic non-small cell lung cancer who have been receiving molecular targeted therapy, including immune checkpoint inhibitor, and have tumor shrinkage with the agent.

Exclusion Criteria:

* Any concurrent and/or other active malignancy that has required treatment within 3 years
* Patients with mixed small cell histology
* Life expectancy less than 3 months
* Insufficient tissue for NGS test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inoperable non-small cell lung cancer with two cohorts as below:
  1. Cohort A: Patients who are diagnosed with metastatic/recurrent non-small cell lung cancer and planned to receive first line chemotherapy
  2. Cohort B: Patients with recurrent/metastatic non-small cell lung cancer who have been receiving molecular targeted therapy, including immune checkpoint inhibitor, and have tumor shrinkage with the agent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Concordance rate | an average of one year
  Concordance rate of genomic change between tumor tissue (FFPE) and ctDNA

SECONDARY OUTCOMES:
Overall survival | an average of one year
  To evaluate prognostic role of ctDNA concentration in NSCLC
Frequency of actionable genomic change | an average of one year
  To determine the frequency of actionable oncogenic genes in NSCLC
Overall survival by treatment | an average of one year
  To evaluate the survival of patients treated with genotype-directed therapy in daily practice

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided